CLINICAL TRIAL: NCT00700219
Title: Development of a Non-invasive Test to Detect Intra-amniotic Infection and Predict Preterm Birth in Women Presenting With Preterm Labor and and Intact Amniotic Membranes
Brief Title: Non-invasive Test to Detect Intra-amniotic Infection in Women With Preterm Labor and Intact Amniotic Membranes
Acronym: IAI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ProteoGenix, Inc. (Industry)
Collaborators: Obstetrix Medical Group (Industry)
Responsible Party: Durlin Hickok, MD, MPH, ProteoGenix, Inc.
Other Study IDs: PGX01-OBX0006
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2010-07

CONDITIONS: Intra-amniotic Infection
Keywords: Preterm Labor; Preterm Birth; Intra-amniotic Infection; Pregnancy; Women
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cervical-vaginal Fluid, Amniotic Fluid, Maternal Serum, Neonatal Cord Blood, Maternal Urine, Placental and Umbilical Cord Tissues
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Women presenting in preterm labor with intact amniotic membranes

SUMMARY:
The purpose of this study is to collect clinical specimens and corresponding clinical data to develop a non-invasive test for detection of intra-amniotic infection and prediction of preterm birth in women and intact amniotic membranes. The specimens collected will be used to develop a specific biomarker panel and algorithm using immunoassays for optimal detection of intra-amniotic infection in women with preterm labor and intact amniotic membranes.

DETAILED DESCRIPTION:
Intra-amniotic infection (IAI) is an acute bacterial infection of the amniotic fluid and intrauterine contents during pregnancy and occurs in 4% to 10% of all deliveries (Newton, ER., 1993. Newton, ER, et al., 1989. Soper, DE, et al., 1989). IAI is an important cause of maternal and neonatal morbidity. Identifying and appropriately treating women with IAI is, therefore, a major obstetrical challenge.

Intrauterine infection may occur early in pregnancy and remain undetected for a prolonged period, thus exposing the fetus to the effects of infection/inflammation for a considerable period. Ideally, an early diagnosis of IAI is important to allow timely treatment and intervention. Unfortunately, the early diagnosis is difficult because the clinical signs and symptoms of IAI may occur late in the course of the infection and are neither sensitive nor specific. Therefore, to avoid a delay in diagnosis a high degree of suspicion and the appropriate use of adjunctive laboratory tests are warranted.

ELIGIBILITY:
Inclusion Criteria:

* Subject is greater than or equal to 18 years of age
* Subject has singleton gestation
* Subject has fetus with gestational age greater than or equal to 22 0/7 weeks and less than or equal to 36 6/7 weeks
* Subject has documented intact amniotic membranes
* Subject's care provider plans to or has performed an amniocentesis procedure
* Subject has had evidence of spontaneous preterm labor as evidenced by documented regular uterine contractions (greater than or equal to four per hour, or if less than 26 weeks gestation, cramping or backache) and one or more of the following:

  1. Progressive cervical change with cervical dilation of greater than or equal to 2 cm
  2. Effacement of greater than or equal to 50%
  3. Cervical length of less than or equal to 30 mm via transvaginal ultrasound
  4. Positive fetal fibronectin test

Exclusion Criteria:

* Subject has documented ruptured amniotic membranes
* Subject has fetus with major fetal anomaly or chromosomal aneuploidy
* Subject has medical indication for preterm birth (e.g. pre-eclampsia)
* Subject is unable to provide written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women presenting to labor and delivery with signs and symptoms of preterm labor and documented intact amntiotic membranes
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Performance of immunoassay panel to detect intra-amniotic infection in target population. | Presentation to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Combs, MD, PhD, Principal Investigator — Obstetrix Medical Group of California
Locations (21):
- United States (21):
  - Banner Desert Memorial Medical Center, Mesa, Arizona
  - Banner Good Samaritan Hospital, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Long Beach Memorial Hospital, Long Beach, California
  - Good Samaritan Hospital, San Jose, California
  - Presbyterian St. Luke's Medical Center, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Norton Downtown, Louisville, Kentucky
  - St. Louis University School of Medicine, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Carolinas Medical Center /Dept. OB/GYN, Charlotte, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Greater Cincinnati Medical Center, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Thomas Jefferson University Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UMCG Dept of OB/GYN, Greenville, South Carolina
  - Swedish Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Combs CA, Garite TJ, Lapidus JA, Lapointe JP, Gravett M, Rael J, Amon E, Baxter JK, Brady K, Clewell W, Eddleman KA, Fortunato S, Franco A, Haas DM, Heyborne K, Hickok DE, How HY, Luthy D, Miller H, Nageotte M, Pereira L, Porreco R, Robilio PA, Simhan H, Sullivan SA, Trofatter K, Westover T; Obstetrix Collaborative Research Network. Detection of microbial invasion of the amniotic cavity by analysis of cervicovaginal proteins in women with preterm labor and intact membranes. Am J Obstet Gynecol. 2015 Apr;212(4):482.e1-482.e12. doi: 10.1016/j.ajog.2015.02.007. Epub 2015 Feb 14. PMID 25687566